CLINICAL TRIAL: NCT00507520
Title: The Effect of Almonds on Coronary Heart Disease Risk Factors: Dose Response Study.
Brief Title: Almond Dose Response Study.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: REB 235U; U of T Protocol #6440
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Last update posted 2007-07-26 (Estimated); Status verified 2007-07

CONDITIONS: Hyperlipidemia; Diet Therapy; Cardiovascular Disease
Keywords: RCT; Almonds; Hyperlipidemia; Blood Lipids
MeSH Terms: conditions — Hyperlipidemias; Cardiovascular Diseases

INTERVENTIONS:
Procedure: Full dose almonds
Procedure: Half dose almonds+half dose muffin
Procedure: Full dose whole wheat muffin

SUMMARY:
To assess the effects of almonds on coronary heart disease (CHD) risk factors (serum lipids, measurements of oxidative stress and nitric oxide production) when added to the diets of subjects with high cholesterol. Also, to assess whether the amount of almonds consumed (i.e. almond dose) decreases CHD risk factors in a dose dependent manner. We hypothesize that since almonds have been shown to reduce serum lipids, we believe they will also increase nitric oxide levels related to their high levels of arginine and reduce markers of oxidative stress related to their content of bioactive phenolics. We anticipate that a dose-dependent relationship will be observed resulting in greater reductions in risk factors for coronary heart disease when greater doses of almonds are consumed.

DETAILED DESCRIPTION:
Previous studies have shown that nuts, specifically almonds, result in an improved coronary heart disease (CHD) lipid risk profile. Part of the reason has been ascribed to their high content of monounsaturated fat. However in a previous study we have done, the almond supplement, in comparison with an olive oil and dairy protein based supplement, still showed a significant reduction in total cholesterol (total-C) and low density lipoprotein cholesterol (LDL-C). We wish to use this paradigm to confirm the lipid lowering effect of almonds, to establish a similar relationship for the apolipoproteins and so add further support for the cardiovascular risk reduction associated with an almond diet. In addition, in view of the relatively high arginine content of almonds, we believe higher levels of nitric oxide (NO) will be produced, as indicated by increased NO in expired air from perfused olfactory mucosa. With this technique, we have found higher levels of NO in preliminary studies of subjects on soy diets. These data would further add to interest in nuts in relation to cardiovascular disease risk reduction. Furthermore, phenolics are present in high concentrations in oil seeds and nuts, and are known to have antioxidant activity. As yet, they do not appear to have been emphasized in relation to almonds. We will therefore determine the effect of feeding almonds on measures of oxidative stress, including oxidized LDL-C, considered to be of direct relevance to CHD; and oxidized DNA, of potential importance to neoplastic transformation and carcinogenesis.

These studies could lead to assessment of postprandial effects of almonds to determine a mechanism, and to studies of cardiovascular effects of almonds including exercise stress tests and measures of vascular reactivity (e.g. forearm blood flow) in conjunction with NO measurements.

Protocol: All subjects underwent three 4-week treatments in a randomized crossover trial.

Background Diet: Subjects were instructed to follow the National Cholesterol Education Program (NCEP) Step 2 dietary guidelines. Nuts, soy and dietary supplements (vitamins, minerals or herbal remedies) were excluded in the background diet during all phases of the study.

Treatments: The three phases were all weight maintaining, self-selected diets: control, full almond and half almond. Almond: Raw almonds were added as supplements to the subject's usual diet. Subjects with calorie needs of 2,400 kcal or greater, assessed by LRC tables, received the full almond supplement (100 g/d, approximately 600 kcal). Subjects requiring between 1,600-2,400 kcal daily received 75% of the full supplement (75 g/d, approximately 450 kcal). Subjects requiring less than 1,600 kcal daily received 50% of the full supplement (50 g/d, approximately 300 kcal). Control: The full control supplement was four 150 kcal muffins. Control supplements was matched with the energy content of the nut supplements; i.e. either 600 kcal/d (4 muffins); 450 kcal/d (3 muffins) or 300 kcal/d (2 muffins). The macronutrient composition of the muffins conformed to an NCEP Step 2 diet with 25% total fat, <7% saturated fat (by use of corn oil as the oil commonly used in healthy baked goods), with 18% protein (the average for our subject population using added skim milk powder), and zero cholesterol. Muffins were made with wheat flour. Half Portion: The Half Portion was matched with the energy content of the other two treatment periods. However on this treatment, half of the energy was derived from almonds and half from the control muffins.

Design: Randomized crossover design.

Duration: The study consisted of three months subject recruitment and selection; three 4-week treatment periods where supplements are provided, and at least two-week washout periods between supplements. (Total duration: approximately 7.5 months per subject).

Study Details: Subjects came after a 12h overnight fast to the Risk Factor Modification Center at St. Michael's Hospital (Toronto) immediately prior to commencement of each study and at weekly intervals during the course of each study period. Prior to the start of the study, subjects were instructed on details of the study diet protocol. They were also asked to maintain a constant level of physical activity throughout the course of the study. At all visits, body weight (in kg) was obtained in indoor clothing, without shoes.

Measurements: Bloods were taken at baseline and at weeks 2 and 4 of each phase. Pulmonary air was collected at baseline and at week 4 of each phase. Diet histories were recorded during the last week of each phase.

Compliance:Compliance was assessed from completed one-week diet records where supplement intake is recorded. Diet records were reviewed by the dietitian with the subject at the end of the week. In addition, uneaten supplements were returned, weighed and noted on the menu plans by the dietitian.

ELIGIBILITY:
Inclusion Criteria:

* Men and post-menopausal women
* LDL-C >4.1 mmol/L at recruitment, aged 40-70, living within a 40 km radius of St. Michael's Hospital.

Exclusion Criteria:

* Lipid lowering medications, clinical or biochemical evidence of diabetes, renal or hepatic disease, body mass index (BMI) >32 kg/m2, antibiotic use within the last three months, hormone replacement therapy, smoking or significant alcohol intake (> 1 drink/d) or triglyceride level >4.0 mmol/L.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 1999-12; Study Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
Lipids: Total Cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, apolipoproteins B and AI
Glycemic control: Glucose, insulin, C-peptide (blood and urine).

SECONDARY OUTCOMES:
Clotting Factors: fibrinogen, tissue plasminogen activator, plasminogen activator inhibitor, urokinase, factor VII and factor VIII.
Oxidative Stress: Oxidized LDL-C as conjugated dienes in isolated LDL-C fraction, serum carotenoids, vitamin E, vitamin A; 8-hydroxy-2-deoxyguanosine (8-HDG) in isolated blood lymphocytes; malondialdehyde (MDA); urinary isoprostanes.
Nitric Oxide: Pulmonary (expired air) NO measured as a marker of whole body NO production and olfactory epithelial NO production in perfused nasal air.

CONTACTS AND LOCATIONS:
Overall Officials: David JA Jenkins, MD, PhD, Principal Investigator — University of Toronto, St. Michael's Hospital; Cyril WC Kendall, PhD, Study Director — University of Toronto, St. Michael's Hospital
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Jenkins DJ, Kendall CW, Marchie A, Parker TL, Connelly PW, Qian W, Haight JS, Faulkner D, Vidgen E, Lapsley KG, Spiller GA. Dose response of almonds on coronary heart disease risk factors: blood lipids, oxidized low-density lipoproteins, lipoprotein(a), homocysteine, and pulmonary nitric oxide: a randomized, controlled, crossover trial. Circulation. 2002 Sep 10;106(11):1327-32. doi: 10.1161/01.cir.0000028421.91733.20. PMID 12221048
- [Derived] Nishi SK, Kendall CWC, Bazinet RP, Hanley AJ, Comelli EM, Jenkins DJA, Sievenpiper JL. Almond Bioaccessibility in a Randomized Crossover Trial: Is a Calorie a Calorie? Mayo Clin Proc. 2021 Sep;96(9):2386-2397. doi: 10.1016/j.mayocp.2021.01.026. Epub 2021 Apr 11. PMID 33853731